CLINICAL TRIAL: NCT00953485
Title: Clinical Trial of Allogeneic Mesenchymal Stem Cells Transplantation for Primary Sjögren's Syndrome - Phase Ⅰ/Ⅱ
Brief Title: Allogeneic Mesenchymal Stem Cells Transplantation for Primary Sjögren's Syndrome (pSS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, the Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJGLYY002
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Sjogren's Syndrome; Mesenchymal Stem Cells
Keywords: Sjogren's Syndrome; Mesenchymal Stem Cells; Transplantation
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Stem Cells (AlloMSC) — Allogeneic mesenchymal stem cells will be infused intravenously (single dose, 10^6 cells/kg body weight).

SUMMARY:
This study will explore safety and efficacy of allogeneic mesenchymal stem cells transplantation (MSCT) to treat patients with diagnosis of primary Sjögren's Syndrome (pSS) who have been resistant to multiple standard treatments. The underlying hypothesis is that the pSS condition is caused by an abnormal immune homeostasis that can be restored by MSCT.

DETAILED DESCRIPTION:
* To test a new approach using allogeneic derived mesenchymal stem cell based therapy (MSCT) to treat refractory primary Sjögren's Syndrome (pSS)
* To determine the disease-free survival in pSS patients treated with MSCT in terms of disease activity index, pSS serology and salivary gland function
* To assess adverse events of allogeneic MSC transplantation
* To assess the association of disease activity index, pSS serology levels, and saliva flow rate at baseline with disease-free survival

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the international classification criteria (2002) for primary Sjögren's Syndrome, man or woman aged from 15 to 70 years old, Sjögren's Syndrome Disease Activity Index (SSDAI)≥8.
* Stimulated whole saliva flow rate less than 1~6ml/6min.
* Patients must be informed of the investigational nature of this study and give written informed consent in accordance with the institutional and hospital guidelines.
* Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on this trial and for 12 months following treatment. Women of child-bearing potential must have a pregnancy test performed within 72 hours prior to initiation of treatment.

Exclusion Criteria:

* End-stage renal failure.
* Severe cardiopulmonary compromise, or other system failure.
* Active, uncontrolled infections.
* Pregnant or nursing women may not participate due to the possibility of fetal harm or harm to nursing infants from this treatment regimen.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Sjögren's syndrome disease activity index | Monthly

SECONDARY OUTCOMES:
pSS Serology (ANA, dsDNA, SS-A, SS-B) | Monthly
Improvement of salivary gland function (measured as stimulated saliva flow rate) | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Lingyun Sun, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Sun L, Akiyama K, Zhang H, Yamaza T, Hou Y, Zhao S, Xu T, Le A, Shi S. Mesenchymal stem cell transplantation reverses multiorgan dysfunction in systemic lupus erythematosus mice and humans. Stem Cells. 2009 Jun;27(6):1421-32. doi: 10.1002/stem.68. PMID 19489103
- [Background] Liang J, Zhang H, Hua B, Wang H, Wang J, Han Z, Sun L. Allogeneic mesenchymal stem cells transplantation in treatment of multiple sclerosis. Mult Scler. 2009 May;15(5):644-6. doi: 10.1177/1352458509104590. PMID 19389752
- [Background] Zhou K, Zhang H, Jin O, Feng X, Yao G, Hou Y, Sun L. Transplantation of human bone marrow mesenchymal stem cell ameliorates the autoimmune pathogenesis in MRL/lpr mice. Cell Mol Immunol. 2008 Dec;5(6):417-24. doi: 10.1038/cmi.2008.52. PMID 19118507
- [Background] Sun LY, Zhang HY, Feng XB, Hou YY, Lu LW, Fan LM. Abnormality of bone marrow-derived mesenchymal stem cells in patients with systemic lupus erythematosus. Lupus. 2007;16(2):121-8. doi: 10.1177/0961203306075793. PMID 17402368
- [Derived] Xu J, Wang D, Liu D, Fan Z, Zhang H, Liu O, Ding G, Gao R, Zhang C, Ding Y, Bromberg JS, Chen W, Sun L, Wang S. Allogeneic mesenchymal stem cell treatment alleviates experimental and clinical Sjogren syndrome. Blood. 2012 Oct 11;120(15):3142-51. doi: 10.1182/blood-2011-11-391144. Epub 2012 Aug 27. PMID 22927248